CLINICAL TRIAL: NCT02598037
Title: Association Between the Change of the Genes With the Hormones and Food Consumption of Obese
Brief Title: Association Between the Change of the Genes With Hormones and Food Consumption of Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Fernanda Cristina Carvalho Mattos Magno, MSc, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 31573114.1.0000.5257
Record Dates: First submitted 2015-10-31; First posted 2015-11-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Obesity; Polymorphism; Hormones
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FTO gene polymorphism (Other): test meal after fasting for 12 hours
  Interventions: Dietary Supplement: Test meal

INTERVENTIONS:
Dietary Supplement: Test meal — The test meal will contain the following features: 50% carbohydrate, 20% protein and 30% of total fat, and will be admnistrada after drawing blood fasting for 12 hours.

SUMMARY:
Obesity is considered one of the most troubling chronic diseases for public health because of its rapid growth in the population. Many are the causal factors of this epidemic, and in recent years studies suggest the involvement of genetic factors in the etiology of obesity as a risk factor for its development. Polymorphism of the FTO gene is being studied in the past eight years and has been indicated as a predictor of obesity in the population, as well as associations in food intake, raising the possibility of influence in the regulation of hunger and satiety. Accordingly, researchers observed changes in levels of postprandial leptin and ghrelin, which can promote appetite and change the quantity and quality of food intake in subjects with the polymorphism FTO.

DETAILED DESCRIPTION:
Obesity is a chronic disease with high growth in the world population, as well as being a risk factor for the development of other chronic diseases. Additionally, it is known that it is a multifactorial disease and polygenic, making it difficult to control. It is also recognized that some environmental factors, with emphasis on diet, can modulate the expression of certain genes and may help control obesity.

In recent decades, researchers from several countries has been devoted to studies that aim to propose alternatives for the treatment of obesity, emphasizing the regulation of energy balance and changes in lifestyle (diet and exercise), and try to clarify the reason some individuals more susceptible to these factors than other, favoring the body weight gain. These differences may be explained in part, by genetic factors.

The FTO gene has been considered a strong candidate gene for obesity because of its relation to the secretion of ghrelin, an important orexigenic hormone involved in the regulation of food intake, which could open new perspectives for studies of gene-environment interactions in obesity.

Considering the significant increase of obesity in the world population, it is understood that studies assessing environmental factors - particularly diet - and genes and genetic variants associated with obesity - may represent a major breakthrough in understanding the development of this disease, providing tools to propose possible changes in current dietary prescriptions for this population.

Also highlighted the lack of studies on the subject, which makes this proposal is innovative and unprecedented as it aims to evaluate the relationship between the FTO gene polymorphism with ghrelin secretion and food intake in obese.

It is suggested that obese individuals with a polymorphism in the FTO gene present higher serum concentrations of basal ghrelin and postprandial (after-fat meal), and the usual food intake, as well as the postprandial appetite, are associated with the concentrations basal and postprandial ghrelin, respectively. These results may generate data for changes in dietary prescriptions aimed at reducing the secretion and, or sensitivity to the hormone to control energy intake, whereas the individual's genotype can not be changed voluntarily in the current state of the art.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with grade 3 obesity.

Exclusion Criteria:

* Pregnant women, teenagers, elderly, use of corticosteroids, medicines for weight loss, bariatric surgery and affected by chronic diseases, such as hyperthyroidism or hypothyroidism, nephropathy, neuropathy, and inflammatory bowel disease. Also excluded are volunteers who do not fulfill all stages of the study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2014-09; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with or without polymorphism ih genes as determined by PCR | Three hours after the test meal
  Genotyping will be used to separate patients by genotypes.

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values for hormones. | Three hours after the test meal
  The hormonal analysis performed by the luminex method will be performed to evaluate the release of hormones between the genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda CM Magno, MSc, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro - CCS, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennan IM, Luscombe-Marsh ND, Seimon RV, Otto B, Horowitz M, Wishart JM, Feinle-Bisset C. Effects of fat, protein, and carbohydrate and protein load on appetite, plasma cholecystokinin, peptide YY, and ghrelin, and energy intake in lean and obese men. Am J Physiol Gastrointest Liver Physiol. 2012 Jul;303(1):G129-40. doi: 10.1152/ajpgi.00478.2011. Epub 2012 May 3. PMID 22556143
- [Background] Deram S, Villares SM. Genetic variants influencing effectiveness of weight loss strategies. Arq Bras Endocrinol Metabol. 2009 Mar;53(2):129-38. doi: 10.1590/s0004-27302009000200003. PMID 19466204
- [Background] Druce MR, Wren AM, Park AJ, Milton JE, Patterson M, Frost G, Ghatei MA, Small C, Bloom SR. Ghrelin increases food intake in obese as well as lean subjects. Int J Obes (Lond). 2005 Sep;29(9):1130-6. doi: 10.1038/sj.ijo.0803001. PMID 15917842
- [Background] Erdmann J, Topsch R, Lippl F, Gussmann P, Schusdziarra V. Postprandial response of plasma ghrelin levels to various test meals in relation to food intake, plasma insulin, and glucose. J Clin Endocrinol Metab. 2004 Jun;89(6):3048-54. doi: 10.1210/jc.2003-031610. PMID 15181097
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Haupt A, Thamer C, Staiger H, Tschritter O, Kirchhoff K, Machicao F, Haring HU, Stefan N, Fritsche A. Variation in the FTO gene influences food intake but not energy expenditure. Exp Clin Endocrinol Diabetes. 2009 Apr;117(4):194-7. doi: 10.1055/s-0028-1087176. Epub 2008 Dec 3. PMID 19053021
- [Background] Karra E, O'Daly OG, Choudhury AI, Yousseif A, Millership S, Neary MT, Scott WR, Chandarana K, Manning S, Hess ME, Iwakura H, Akamizu T, Millet Q, Gelegen C, Drew ME, Rahman S, Emmanuel JJ, Williams SC, Ruther UU, Bruning JC, Withers DJ, Zelaya FO, Batterham RL. A link between FTO, ghrelin, and impaired brain food-cue responsivity. J Clin Invest. 2013 Aug;123(8):3539-51. doi: 10.1172/JCI44403. Epub 2013 Jul 15. PMID 23867619
- [Background] Loos RJ, Bouchard C. Obesity--is it a genetic disorder? J Intern Med. 2003 Nov;254(5):401-25. doi: 10.1046/j.1365-2796.2003.01242.x. PMID 14535962
- [Background] Chen LP, Thomas EK, Hu SL, Hellstrom I, Hellstrom KE. Human papillomavirus type 16 nucleoprotein E7 is a tumor rejection antigen. Proc Natl Acad Sci U S A. 1991 Jan 1;88(1):110-4. doi: 10.1073/pnas.88.1.110. PMID 1846033
- See also: MANAGING OVERWEIGHT AND OBESITY IN ADULTS: SYSTEMATIC EVIDENCE REVIEW FROM THE OBESITY EXPERT PANEL, 2013 — https://www.nhlbi.nih.gov/health-topics/managing-overweight-obesity-in-adults